CLINICAL TRIAL: NCT05241847
Title: Starzl Network for Excellence in Pediatric Transplantation (SNEPT) Implementation of a QoL Measure in Pediatric Transplant Recipients
Brief Title: Starzl Network Patient Reported Outcomes
Acronym: SPaRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); The Hospital for Sick Children (Other); Emory-Children's Center (Other); Columbia University (Other); Seattle Children's Hospital (Other); University of San Francisco (Other)
Responsible Party: Principal Investigator, George Mazariegos, Professor of Surgery, Chief Pediatric Transplantation, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY21090139; U18HS028380-01 (AHRQ)
Record Dates: First submitted 2022-01-22; First posted 2022-02-16 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Liver Transplant; Complications; Quality of Life; Child Behavior; Adolescent Behavior
Keywords: quality of life
MeSH Terms: conditions — Child Behavior; Adolescent Behavior

STUDY DESIGN:
Intervention Model Description: Single arm interventional trial with use of the RTC mobile application representing the intervention of interest
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pediatric liver transplant recipients (Experimental): As this is a single arm trial, all eligible liver transplant recipients and their caregivers will be enrolled in this arm.
  Eligible participants are children who received a liver transplant at least 1 year prior to enrollment at a participating SNEPT center and continue to receive their post-transplant care at that center.
  Interventions: Behavioral: PeLTQL delivery via electronic means

INTERVENTIONS:
Behavioral: PeLTQL delivery via electronic means — Delivery of PeLTQL scoring information to clinicians via electronic means.
  Other Names: Real Time Clinic mobile application

SUMMARY:
This study uses a smartphone application/web interface (RealTime Clinic; RTC) to collect patient and parent reports of a pediatric liver transplant recipient's quality of life (QOL), and examines the extent to which QOL evaluations can be integrated into care with the help of the application. The QOL measure that is used in this study is the Pediatric Liver Transplant Quality of Life (PeLTQL) questionnaire. Utilization, effectiveness, and efficiency data are evaluated.

Hypotheses are fully described in the protocol. The primary hypothesis is that 80% of recruited child-proxy dyads will have at least one RTC-enabled PeLTQL score at 12 months. Other hypotheses look at implementation metrics and patient outcomes.

DETAILED DESCRIPTION:
Despite evidence supporting the benefits of QOL assessments and the availability of many QOL assessment instruments, the integration of these instruments into clinical practice has not yet become standard of care.

The Pediatric Liver Transplant Quality of Life (PeLTQL), the study measure, is a condition-specific 26-item questionnaire; the investigators will be evaluating both total scores as well as subdomain scores and, importantly, discrepancies between child and parent reports of the child's QOL.

The Electronic Platform: Real-Time Clinic (RTC). The platform will furnish providers with the total scores, subscale scores, thresholds ("met" vs. "not met"), discrepancy scores, and any question that has scores which may concern the clinician/clinical team.

This information will be available before the clinic visit and can guide and inform discussion and problem-solving between patient and clinical team. The study does not standardize the response to the results and will not suggest a preferred way of action. Interpretation of the results, as well as actions related to them are completely left to clinician's discretion.

The setting of this study - the Starzl Network for Excellence in Pediatric Transplantation (SNEPT Centers). SNEPT is a learning healthcare network that was established in 2018 to accelerate improvement in transplant outcomes by incorporating innovation, technology and the patient voice to address gaps in care that were identified by the collaborative transplant centers and family representatives.

Study Aims

The primary aim is successful implementation of the RTC app-based tool to obtain PeLTQL scores from pediatric liver transplant recipients and their parents or caregivers.

The investigators also aim to assess the usability, impact, and ease of use (both for clinicians and patients/families) of the RTC platform and app-based version of the PeLTQL. The investigators will evaluate clinicians' subjective views on the platforms' ease of use, their time spent evaluating results, both in clinic and before patient visits, as well as the app's impact on back-end clinic workflow.

Impact on patient outcomes will be evaluated using pre-post comparisons on adherence (determined by the objective medication level variability index, MLVI) as well as on the PeLTQL.

ELIGIBILITY:
Inclusion Criteria:

The patient must meet all of below criteria to be eligible for enrollment in the study:

1. The patient is > 8 at enrollment and < 20 years of age at 2 year post enrollment.
2. The patient received a liver transplantation at least 1 year prior to enrollment.
3. The patient and parent/ guardian have internet access either through a smartphone, tablet or computer.
4. The patient and at least one guardian speaks English or Spanish at a level that allows them to understand the study procedures and consent to the study.

Exclusion Criteria:

None of the following may be present if the patient is to be eligible for enrollment in the study:

1. The patient is expected to transition to another service (e.g., adult clinic, another hospital) in the year following enrollment.
2. The guardian or patient (in a developmentally-appropriate manner) do not understand the study procedures. This will be verified by asking both guardian and adolescent to repeat the study procedures.

Ages: 8 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Implementation metric | 12 months
  The proportion of participants who complete the Pediatric Liver Transplant Quality of Life (PeLTQL) measure (either parent or child), at least once

SECONDARY OUTCOMES:
Patient baseline quality of life (child report on PeLTQL) | Time of enrollment
  PeLTQL = Pediatric Liver Transplant Quality of Life questionnaire. Range of scores (after transformation), range (0-100) Higher score = Better QoL
Patient quality of life (child report on PeLTQL) | 12 months post-enrollment
  PeLTQL = Pediatric Liver Transplant Quality of Life questionnaire. Range of scores (after transformation), range (0-100) Higher score = Better QoL
Proxy report of child's quality of life using PeLTQL | Time of enrollment
  PeLTQL = Pediatric Liver Transplant Quality of Life questionnaire. Range of scores (after transformation), range (0-100) Higher score = Better QoL
Proxy report of child's quality of life using PeLTQL | 12 months post-enrollment
  PeLTQL = Pediatric Liver Transplant Quality of Life questionnaire. Range of scores (after transformation), range (0-100) Higher score = Better QoL
Medication level variability index (MLVI) | Calculated for year following implementation (12 month period following enrollment)
  Degree of fluctuation in immunosuppressant medication levels. Higher MLVI =worse adherence to medication.
PeLTQL discrepancy score | First administration of PeLTQL in year 1
  The discrepancy score is defined as the parent score minus the child's score on the PELTQL. PeLTQL = Pediatric Liver Transplant Quality of Life questionnaire
PeLTQL discrepancy score | Second administration of PeLTQL within 24 months
  The discrepancy score is defined as the parent score minus the child's score on the PELTQL. PeLTQL = Pediatric Liver Transplant Quality of Life questionnaire
Implementation metric | 18 months
  Percentage of patient-proxy dyads (amongst all enrolled) who completed the PeLTQL at least once.
Implementation metric | 24 months
  Percentage of participating parent-child dyads (amongst all dyads) in which both the parent and the child completed one or more questionnaires during the study period.

OTHER OUTCOMES:
Rejection | 24 months
  Incidence of rejection of the transplanted liver

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Shemesh, MD, Principal Investigator — Icahn School of Medicine at Mt. Sinai; George Mazariegos, MD, Principal Investigator — University of Pittsburgh
Locations (7):
- United States (6):
  - UCSF Benioff Children's Hospital, Oakland, California
  - Emory Children's, Atlanta, Georgia
  - Columbia University Children's, New York, New York
  - Mt. Sinai, New York, New York
  - UPMC Children's, Pittsburgh, Pennsylvania
  - Seattle Children's, Seattle, Washington
- Toronto Sick Kids, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ng V, Nicholas D, Dhawan A, Yazigi N, Ee L, Stormon M, Gilmour S, Schreiber R, Taylor R, Otley A; PeLTQL study group. Development and validation of the pediatric liver transplantation quality of life: a disease-specific quality of life measure for pediatric liver transplant recipients. J Pediatr. 2014 Sep;165(3):547-55.e7. doi: 10.1016/j.jpeds.2014.05.024. Epub 2014 Jun 26. PMID 24976329
- See also: Starzl Network Main Website — http://starzlnetwork.org/